CLINICAL TRIAL: NCT03824496
Title: Measuring Cardiac Head Impulse to Detect Acute Large Vessel Ischemic Stroke
Brief Title: Head Pulse for Ischemic Stroke Detection
Acronym: EPISODE
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 17-21846
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected acute stroke: Any patient with suspected acute stroke triggering a "stroke code" and had a brain imaging angiogram
  Interventions: Diagnostic Test: Cranial Accelerometry Measurement

INTERVENTIONS:
Diagnostic Test: Cranial Accelerometry Measurement — Measuring the HeadPulse using cranial accelerometry

SUMMARY:
Accurate diagnosis of stroke due to large vessel occlusion (LVO) is an essential step in providing acute stroke care to a community. The gold-standard for diagnosis LVO is brain imaging, which is impractical in the pre-hospital setting. A non-invasive method to detect LVO is needed. Using highly sensitive accelerometers, one can measure the "HeadPulse"- tiny forces exerted on the skull from the cardiac contraction. This study tests the hypothesis that LVO alters the HeadPulse characteristically. Analysis of these data along with the subjects vascular status (LVO vs. non-LVO as measured by CT angiography) will be used to create a model that can predict LVO status in suspect stroke subjects.

DETAILED DESCRIPTION:
Large vessel occlusion (LVO) ischemic stroke is a treatable disease at specialized centers. Clinical outcomes of patients with LVO is time-dependent. To maximize clinical benefit of thrombectomy, stroke systems of care need accurate methods to triage patients with LVO to comprehensive stroke centers or thrombectomy ready centers rather than closer primary stroke centers.

EPISODE will evaluate whether measurements of the HeadPulse can predict the presence or absence of LVO based on recordings from a consecutive series of patients undergoing CTA for suspected stroke. Recordings from patients pre- and post-thrombectomy will also be compared to investigate whether a systematic change in cranial forces exists during LVO.

ELIGIBILITY:
Inclusion Criteria:

* Suspected acute stroke
* CTA or MRA performed

Exclusion Criteria:

* Any patient in whom obtaining a non-invasive recording is judged by the treating team to interfere with clinical assessment or treatment of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been evaluated by a medical professional who feels the subject may be experiencing an acute stroke and has triggered the acute stroke algorithm within the medical center.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2019-08-18 (Actual)

PRIMARY OUTCOMES:
Cranial accelerometry model | Through study completion, likely 2 years
  Difference in cranial accelerometry waveform analysis in LVO vs. non-LVO subjects

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No